CLINICAL TRIAL: NCT00002192
Title: Tolerance, Safety, and Activity of Rifapentine Alone and in Combination Therapy in AIDS Patients With Mycobacterium Avium Complex Bacteremia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anderson Clinical Research (Industry)
Collaborators: Hoechst Marion Roussel (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 275A; 000473PR0018; 96ACR-HMD1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Antitubercular Agents; Azithromycin; Clarithromycin; Bacteremia; rifapentine
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Bacteremia | interventions — rifapentine; Ethambutol; Clarithromycin; Azithromycin

INTERVENTIONS:
Drug: Rifapentine
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Azithromycin

SUMMARY:
To determine the antimicrobial activity and tolerability of rifapentine alone and in combination therapy in patients with AIDS and disseminated Mycobacterium avium complex (MAC) bacteremia. To determine the pharmacokinetics of rifapentine and its metabolite, 25-desacetyl, alone and in combination therapy. To determine the pharmacokinetics of azithromycin and clarithromycin (and its 14-OH metabolite) in combination therapy.

DETAILED DESCRIPTION:
This open-label, sequential study is conducted in two parts: a monotherapy phase and a combination treatment phase.

In the monotherapy phase sequential 3-patient cohorts receive 1 of 3 doses of rifapentine monotherapy.

In the combination treatment phase, 12 patients each are randomized to one of three arms:

Arm I: Rifapentine (assigned dose level based on monotherapy phase) plus azithromycin.

Arm II: Rifapentine (assigned dose level) plus clarithromycin. Arm III: Rifapentine (assigned dose level) plus ethambutol.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented positive HIV serology status.
* Documented AIDS.
* Positive blood culture for MAC from the study-designated microbiology laboratory. NOTE:
* Patients with presumed MAC bacteremia, as evidenced by positive blood, bone marrow, or liver biopsy culture analyzed locally, may be enrolled pending confirmation.
* Minimum of two MAC-associated symptoms, defined as >= grade 1 fever; > grade 1 night sweats, fatigue, diarrhea, abdominal pain, or anorexia; or weight loss > 5% reported within 4 weeks prior to study entry.
* Life expectancy of at least 3 months.

Prior Medication:

Allowed:

MAC prophylaxis with medications other than study drugs (5-day washout period required).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Pulmonary tuberculosis.
* Infections requiring the use of disallowed medications.
* Serious diseases that introduce undue risks for adverse reactions to study medication.

Concurrent Medication:

Excluded:

* Terfenadine.
* Treatment for pulmonary TB.
* Study drugs from an outside source.
* Medications with anti-MAC activity (i.e., amikacin, ciprofloxacin, clofazimine, rifampin, and rifabutin).

Patients with the following prior conditions are excluded:

* History of hypersensitivity to rifabutin, rifampin, clarithromycin, erythromycin, azithromycin, or ethambutol.
* Previous episode of uveitis.

Prior Medication:

Excluded:

* Prophylactic treatment for MAC with rifabutin or any of the study medications.
* Azithromycin within the 3 weeks prior to randomization.
* Any investigational drug during the 4 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hampton Roads Med Specialists, Hampton, Virginia, United States